CLINICAL TRIAL: NCT07269483
Title: Sunrise in Obstructive Sleep Apnoea Study (SOSA) A Comparison of the Sunrise Mandibular Movement Monitoring Device With Overnight Oximetry and WatchPAT in the Diagnosis and Management of Obstructive Sleep Apnoea.
Brief Title: A Study Assessing Adult Patients Referred to an NHS Sleep Service With Suspected Obstructive Sleep Apnoea. This Study Aims to Compare the Sunrise Wearable Diagnostic Device Performance and Potential Inclusion in a NHS Diagnostic Pathway With Oximetry and WatchPAT Which Are Currently Used.
Acronym: SOSA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Virginia Hawkins (Other)
Collaborators: University Hospitals Bristol and Weston NHS Foundation Trust (Other)
Responsible Party: Sponsor-Investigator, Virginia Hawkins, Chief Investigator - Senior Lecturer, Manchester Metropolitan University
Organization: Manchester Metropolitan University (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: REC reference: 25/NW/0102
Record Dates: First submitted 2025-11-25; First posted 2025-12-08 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-11

CONDITIONS: Obstructive Sleep Apnoea (OSA)
Keywords: Obstructive Sleep Apnoea; Home-testing devices for Obstructive Sleep Apnoea; sleep-disordered breathing; Excessive daytime sleepiness; Sunrise device; WatchPAT 300; Overnight oximetry; wearable sleep diagnostic device; Home sleep study; mandibular movement monitoring; diagnostic accuracy study; single-centre study; digital health technology; patient experience; patient feedback; NHS innovation; waiting list reduction; machine learning in sleep medicine; Home-testing devices for diagnosing obstructive sleep apnoea hypopnoea syndrome NICE guidance 2024; diagnostic pathway efficiency; Obstructive Sleep Apnoea Hypopnoea syndrome; patient reported outcomes; cost effectiveness
MeSH Terms: conditions — Sleep Apnea, Obstructive; Sleep Apnea Syndromes; Disorders of Excessive Somnolence | interventions — Oximetry

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: * The Principal Investigator (PI) and Clinical fellow will be blinded to the CRF after visit 1 to help ensure unbias analysis and triaging of Sunrise results. The database manager will complete the CRF after this point and update the study spreadsheet with the results.
  * Sunrise results will be triaged by the PI and the clinical fellow. Both will be blinded to the oximetry and WatchPAT 300 triage outcome.
  * The unblinded investigators within UHBW will be the co-investigator and the trial database manager.
  * The PI and clinical fellow who will be triaging the Sunrise result will be blinded to the results of the WatchPAT 300 or oximetry result, and the clinical management decision made based on the WatchPAT 300 or oximetry result.
  Once data collection and triaging has finished, the oximetry and WatchPAT 300 result and the clinical management decision made on those results will be made available to the PI to analyse the study outcomes.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- WatchPAT 300 (Experimental): WatchPAT 300 and Sunrise
  Interventions: Diagnostic Test: WatchPAT 300; Diagnostic Test: Sunrise
- Oximetry (Experimental): Oximetry and Sunrise
  Interventions: Diagnostic Test: Oximetry; Diagnostic Test: Sunrise

INTERVENTIONS:
Diagnostic Test: WatchPAT 300 — Participants will use the Sunrise diagnostic device simultaneously with their NHS sleep study - WatchPAT.
  Arms: WatchPAT 300
Diagnostic Test: Oximetry — Participants will use the Sunrise diagnostic device simultaneously with their NHS sleep study - oximetry.
  Arms: Oximetry
Diagnostic Test: Sunrise — Patients will use the Sunrise device which is a submandibular wearable for overnight sleep studies

SUMMARY:
The goal of this clinical trial is to evaluate whether the Sunrise device (that measure small jaw movements) can improve the diagnosis and management of Obstructive Sleep Apnoea (OSA) in adults (≥ 18 years) referred to a Sleep Clinic.

The main question it aims to answer are:

- Does Sunrise lead to a higher proportion of definitive management decisions (initiate OSA treatment, discharge from the sleep clinic service, additional diagnostic testing required or a clinic appointment) compared to current screening practices, which includes either overnight oximetry or use of a wearable device called WatchPAT 300?

Researchers will compare Sunrise results with oximetry and WatchPAT 300 outcomes to see if Sunrise improves diagnostic efficiency, reduces time to a diagnosis or clinical decision and enhances patient experience.

Participants will:

* Follow the standard clinical pathway (oximetry or WatchPAT 300)
* Use the Sunrise device simultaneously for one night with their usual test
* Complete a patient feedback questionnaire on ease of use and experience
* Return all equipment two days later, Sunrise results will not affect their clinical care and will be used for the study only

DETAILED DESCRIPTION:
The study was designed to answer whether Sunrise can be used as an alternative sleep diagnostic test in an existing clinical pathway. Previous research has validated the device against Gold Standard testing - full polysomnography and polygraphy. Previous research has deemed the Sunrise device demonstrated a 92% accuracy when comparing full polysomnography to Sunrise and another study demonstrated 88-100% accuracy depending on OSA severity when tested in a patients home instead of an in patient sleep laboratory. Future research suggested evaluating the Sunrise device in a variety of care pathways and suggested patient experience to be considered.

The NICE guidance published 19/12/24, reviewing novel home testing devices for OSA highlights gaps in the research, including the need to review the accuracy in home testing devices at diagnosing and assessing OSA severity in patients with brown or black skin. University Hospitals Bristol and Weston NHS Foundation Trust sleep department receives referrals from all ethnic groups and we plan to include a range of ethnicity in our study.

This study aims to address research gaps by comparing the performance of Sunrise with oximetry and WatchPAT in the assessment of patients with suspected OSA to consider whether it could be incorporated into a standard diagnostic pathway. This will be done in an existing clinical service along side the current clinical care pathway, a range of ethnicity being referred into the service will be screened for recruitment. A patient feedback questionnaire will be issued to the patient on the usability of Sunrise device. There are currently no published studies reviewing Sunrise in a clinical pathway or comparing against diagnostic tests other than polygraphy or full polysomnography.

If the hypothesis is proven, Sunrise has the advantage of requiring no reporting time and can be conveniently posted to patients, and is therefore potentially a viable alternative test for the diagnosis of OSA, speeding up the patient pathway and reducing waiting times. Nationally, waiting sleeps for sleep diagnostic testing is increasing and services are unable to keep up with demand, if the hypothesis is proven, the Sunrise device could be implemented nationally and other sleep services may benefit from this research. This study could also address patient feedback and complaints by avoiding attending the department and subsequently improve patient experience.

This research is being conducted as part of the Principal Investigators HSST doctorate. Methodology training has been provided through planned lecture material delivered by MMU, competing the Good Clinical Practice certificate and competing additional learning through the Research Integrity Training certificate through MMU.

The principle research question is: How does Sunrise compare to overnight oximetry and WatchPAT 300 for diagnosing and managing Obstructive Sleep Apnoea within an adult sleep clinical pathway? The study success will be based on how does Sunrise, a novel device compare in the ability to conclude a clinical management decision against standard and well established diagnostic devices in the NHS sleep service.

The study aims to recruit 100 participants from University Hospitals Bristol NHS Foundation Trust (Bristol Royal Infirmary Hospital) sleep department. The study plans to recruit 5-6 patients per week over 16-20 weeks. This has been calculated based on current referral numbers and staff resources for the study. Patients will be identified by the Principal Investigator and the Clinical Fellow reading the patient referral letters into the service and screening against the inclusion / exclusion criteria. Patients will be sent via post a covering letter and Patient Information sheet.

The study design and research questions ensures participation in the study does not delay patient care or treatment.

Inclusion / exclusion criteria Access to a smartphone is required as the Sunrise device relies on the Sunrise app to transfer the patient's report to the sleep department. This may exclude eligible patients without a smartphone or access to WiFi/ internet data.

UHBW does have patient WiFi which patients can access when they collect and return the equipment. Exclusion criteria include co-morbidities or other sleep disorders that could affect the primary outcome, as well as patients with beards, as this may impact device placement and accuracy. In-patients are excluded due to different care pathways and potential unknown co-morbidities. Easy to follow instructions with pictures and videos for Sunrise device use have been designed to be as inclusive as possible.

The Principal Investigator, Clinical Fellow or Co-Investigator will assess whether patients referred to the service meet inclusion / exclusion criteria by reviewing referral letters for the assessment of OSA and patient demographics on their electronic patient record at UHBW. The Principal Investigator, Clinical Fellow and Co-investigator are clinical members of staff employed by UHBW Trust, already have access to the patient electronic record and are involved in the triaging process and part of the existing clinical care team. No additional screening is required beyond meeting the inclusion/exclusion criteria.

Telephone call:

Potential participants will initially be approached by the Principal Investigator or Clinical Fellow who is part of their normal clinical care team via telephone after screening their referral letter and electronic medical records. The patient will have previously been sent the Patient Information Sheet and will have the ability to ask further questions. If the patient expresses interest in participating, they will be recruited and sign written consent for the study when they attend the department to collect their NHS diagnostic equipment.

Visit 1:

Participants attend the department and meet with the Principle Investigator, Clinical Fellow, Database manager or coinvestigator.

Participation in the study will be discussed again giving the patient the opportunity to ask questions. If the patient agrees to enrol, they will complete the consent paperwork. All enrolled participants will have demographics measured at the appointment where equipment is collected. There are no additional screening tests than the patients existing clinical pathway. Tests include height, weight, Body Mass Index and collar size. Sex, age and ethnicity will be recorded from the medical records and confirmed with the participant. The current clinical pathway triages patient referrals to oximetry or WatchPAT based on age and clinical history.

Patients will leave the department with oximetry and Sunrise or WatchPAT and Sunrise to use for 1 night at the same time in their own home. Patients are issued the new patient questionnaire and an Epworth Sleepiness Score questionnaire and oximetry or WatchPAT instructions as part of their clinical pathway and will be issued a Sunrise patient feedback questionnaire and Sunrise instructions as part of the study. The participants have an appointment two days later to return the equipment which is booked as part of their clinical pathway. No additional appointments or hospital visits are required of the patient participates in the study. Participants will be told their participant number e.g. 001, 002 to input on their Sunrise feedback questionnaire to ensure there is no identifiable information.

Visit 2:

The participant returns the diagnostic equipment to the department and will have the opportunity to speak to the Principal Investigator, Clinical Fellow or database manager if they have any questions or concerns or if there were any issues completing the questionnaires. The patient exits the study at this point and continues their clinical pathway. If the patient was unable to complete the electronic Sunrise patient feedback questionnaire they will be offered a paper version of the questionnaire.

The patient exists the study after visit two and will continue on the clinical care pathway.

Follow up:

There is no patient follow up as part of the study as they will continue the clinical pathway and receive a management decision based on the oximetry or WatchPAT results. Patients will have the option to be informed of the study results by letter once recruitment has finished and results analysed.

The study has been designed with minimal risk and burden to the patient as the study has been designed in line with the existing clinical pathway. This has ensured patients do not require to attend the department for additional visits.

The patient will be required to use the Sunrise device in addition to the oximetry or WatchPAT device which they would be using as part of their existing clinical pathway. The additional burden would be using the Sunrise device at the same time as the oximetry or WatchPAT so two diagnostic studies would be performed simultaneously. The Sunrise device is non-invasive and sticks on the patients chin area. The patient will also be required to complete a Sunrise patient feedback questionnaire in addition to their clinical pathway. To minimise the burden this is accessible via a Quick Reference (QR) image or a paper version can be available.

This research will potentially improve patient experience if the Sunrise device is equivalent to WatchPAT or superior to oximetry in reaching a management decision for Obstructive Sleep Apnoea diagnosis. This could reduce the number of appointments or diagnostic tests patients need to reach a management decision. The Sunrise device has the ability to be posted to patients which would reduce the need for some patients to book time off work, travel to a city centre hospital where there is a clean air zone charge. The device will not be posted to patients as part of this study as patients need to come in to the department to collect the oximetry or WatchPAT device and complete complete consent paperwork for the study. If the hypothesis is proven, the Sunrise device could reduce the patient pathway time from referral to treatment as the Sunrise device auto analyses results and does not require manual analysis. Currently the WatchPAT requires manual analysis which increases the patient pathway as it is dependant on qualified staff availability and training to analyse the results. Oximetry and WatchPAT results are worn on the patient wrist with a finger probe which can fall off the patients finger while they are sleeping. The Sunrise device is smaller and fits on the patients chin, we will review in the patient feedback patients experience with the Sunrise device and their overall preference between the three devices.

Once the patient has returned the diagnostic equipment, they will exit the study but continue on the existing clinical pathway. Participating in the study does not affect their clinical management as the Sunrise results will be triaged to plan a hypothetical management plan which will be compared to their management plan from their oximetry or WatchPAT results. Patients will be notified of the study outcome upon request once data analysis has been completed.

ELIGIBILITY:
Inclusion Criteria:

* • Adults (aged ≥18 years old) referred with suspected Obstructive Sleep Apnoea

  * Patient has capacity to provide informed consent
  * Patient has access to a smartphone with Bluetooth and WiFi or internet data to download the Sunrise app and to transmit the Sunrise results to the Sunrise portal. UHBW Trust Wi-Fi available to the patient at equipment collection and return if needed.
  * Willing and able to comply with the study-specific procedures
  * Ability to read and comprehend English or understand simple device user instructions with guided pictures in English.

Exclusion Criteria:

* • Suspected diagnosis of a sleep disorder other than OSA (including central sleep apnoea, parasomnias, narcolepsy, idiopathic hypersomnia)

  * Suspected chronic hypercapnic respiratory failure (history of acute hypercapnic respiratory failure, raised CO2 or serum bicarbonate)
  * Patients with unstable cardiovascular disease or non-arteritic anterior ischaemic optic neuropathy
  * Patients with beards who are unwilling to shave the area below their lip (the soul patch)
  * Patients with conditions affecting the rotation of the condyle in the temporo-mandibular joint
  * Unable to consent or lacks capacity to provide informed consent
  * In-patient referrals
  * Unwilling or unable to comply with the study-specific procedures.
  * Patients who have requested in their medical notes not to be involved in research or not to receive digital communication

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-07-28 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
The proportion of patients for which a definitive management decision can be made when tested with Sunrise will be determined and compared to that of oximetry and WatchPAT 300. | • Patients recruited into the study will be issued the Sunrise device to use simultaneously for one night with oximetry or WatchPAT 300. • Patient exits the study when both devices are returned. • Sunrise results will be triaged by the PI and fellow
  * The Principal Investigator (PI) will be blinded to the CRF after visit 1 to help ensure unbias analysis and triaging of Sunrise results. The database manager will complete the CRF after this point and update the study spreadsheet with the results.
  * Patients will return the Sunrise device the same time as their oximetry or WatchPAT 300.
  * Patient exits the study at this point. No further study requirements from the patient.
  * Sunrise results will be triaged by the PI and the clinical fellow. Both will be blinded to the oximetry and WatchPAT 300 triage outcome.
  * Hypothetical management plan following Sunrise Triage i) CPAP set up; ii) further diagnostic testing or iii) discharge from sleep service) iv) clinic appointment for further discussion.
  * The patient referral letter and new patient questionnaire will be consulted after Sunrise data hypothetical managements are determined, to compare the patient's clinical pathway following current practice and a CRF completed.

CONTACTS AND LOCATIONS:
Overall Officials: Virginia Hawkins, BSc, Study Chair — Manchester Metropolitan University
Locations (1):
- University Hospitals Bristol and Weston NHS Foundation Trust, Bristol, South West, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared outside of this study.

REFERENCES:
- [Background] Moffa A, Giorgi L, Carnuccio L, Mangino C, Lugo R, Baptista P, Casale M. New diagnostic tools to screen and assess a still too underestimated disease: the role of the wrist-worn peripheral arterial tonometry device-a systematic review. Sleep Breath. 2023 Jun;27(3):817-828. doi: 10.1007/s11325-022-02700-4. Epub 2022 Aug 29. PMID 36036338
- [Background] Martinot JB, Le-Dong NN, Cuthbert V, Denison S, Borel JC, Gozal D, Pepin JL. Respiratory Mandibular Movement Signals Reliably Identify Obstructive Hypopnea Events During Sleep. Front Neurol. 2019 Aug 13;10:828. doi: 10.3389/fneur.2019.00828. eCollection 2019. PMID 31456731
- [Background] Martinot JB, Cuthbert V, Le-Dong NN, Coumans N, De Marneffe D, Letesson C, Pepin JL, Gozal D. Clinical validation of a mandibular movement signal based system for the diagnosis of pediatric sleep apnea. Pediatr Pulmonol. 2022 Aug;57(8):1904-1913. doi: 10.1002/ppul.25320. Epub 2021 Mar 1. PMID 33647188
- [Background] Martinot JB, Borel JC, Cuthbert V, Guenard HJ, Denison S, Silkoff PE, Gozal D, Pepin JL. Mandibular position and movements: Suitability for diagnosis of sleep apnoea. Respirology. 2017 Apr;22(3):567-574. doi: 10.1111/resp.12929. Epub 2016 Nov 6. PMID 28225162
- [Background] Martinot JB, Senny F, Denison S, Cuthbert V, Gueulette E, Guenard H, Pepin JL. Mandibular movements identify respiratory effort in pediatric obstructive sleep apnea. J Clin Sleep Med. 2015 Apr 15;11(5):567-74. doi: 10.5664/jcsm.4706. PMID 25766710
- [Background] Kelly JL, Ben Messaoud R, Joyeux-Faure M, Terrail R, Tamisier R, Martinot JB, Le-Dong NN, Morrell MJ, Pepin JL. Diagnosis of Sleep Apnoea Using a Mandibular Monitor and Machine Learning Analysis: One-Night Agreement Compared to in-Home Polysomnography. Front Neurosci. 2022 Mar 15;16:726880. doi: 10.3389/fnins.2022.726880. eCollection 2022. PMID 35368281
- [Background] Pepin JL, Letesson C, Le-Dong NN, Dedave A, Denison S, Cuthbert V, Martinot JB, Gozal D. Assessment of Mandibular Movement Monitoring With Machine Learning Analysis for the Diagnosis of Obstructive Sleep Apnea. JAMA Netw Open. 2020 Jan 3;3(1):e1919657. doi: 10.1001/jamanetworkopen.2019.19657. PMID 31968116
- See also: Nice Guidelines: Home-testing devices for diagnosing obstructive sleep apnoea hypopnoea syndrome Diagnostics guidance Reference number:DG62 Published: 19 December 2024 — https://www.nice.org.uk/guidance/dg62
- See also: Nice Guidance: Obstructive sleep apnoea/hypopnoea syndrome and obesity hypoventilation syndrome in over 16s (NICE guideline NG 202). — https://www.nice.org.uk/guidance/ng202
- See also: Sunrise website — https://row.hellosunrise.com/pages/landing-us

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2025-04-24): https://cdn.clinicaltrials.gov/large-docs/83/NCT07269483/Prot_SAP_ICF_001.pdf